CLINICAL TRIAL: NCT00057122
Title: Novel TB Prevention Regimens for HIV-Infected Adults
Brief Title: Tuberculosis Prevention for HIV Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Richard Chaisson, Director, Center for TB Research, National Institute of Allergy and Infectious Diseases (NIAID)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01AI048526-01A1 (NIH); 5R01AI048526-02 (NIH)
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Preventive therapy
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Isoniazid; rifapentine; Rifampin

ARMS (4):
- 1 (Active Comparator)
  Interventions: Drug: Isoniazid; Drug: Rifapentine
- 2 (Active Comparator)
  Interventions: Drug: Isoniazid; Drug: Rifampin
- 3 (Active Comparator)
  Interventions: Drug: Isoniazid
- 4 (Active Comparator)
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — 300mg
Drug: Rifapentine — Rifapentine 900 mg
  Arms: 1
Drug: Rifampin — Rifampin 600 mg
  Arms: 2

SUMMARY:
This study compares three different tuberculosis (TB) prevention regimens against the standard regimen of 6 months of isoniazid. It is being conducted in Soweto, South Africa. People who are HIV positive and have a positive tuberculin skin test without signs of active tuberculosis may join.

DETAILED DESCRIPTION:
AIDS is the leading cause of death in sub-Saharan Africa, and TB is the leading cause of death in patients with AIDS on that continent. Preventive therapy for HIV infected people with latent TB infection is important to reduce the risk of progression to active TB. Although preventive TB therapy is generally recommended throughout the Western world for people with HIV, it is not routinely advocated or provided to patients in developing countries. Six months of self-supervised INH is the gold standard of preventive TB therapy. Newer preventive regimens with a shorter duration of treatment and intermittent dosing could improve compliance and permit treatment supervision through dosing observation. This study will compare the standard INH regimen with two new regimens: rifapentine and INH observed once weekly for 12 weeks and rifampin and INH observed twice weekly for 12 weeks.

Patients will be interviewed to identify risk factors for TB and symptoms of active TB. A physical examination and chest radiograph will be performed on all potential patients to identify and exclude all active TB cases (these patients will be referred for appropriate treatment of their infection).

Patients who meet the inclusion criteria will be randomized to one of the following treatment arms: rifapentine/INH for 12 weeks, observed weekly; rifampin/INH for 12 weeks, observed twice weekly; INH for 6 months, self-supervised; or continuous INH, self-supervised. Patients randomized to the two self-administered INH arms will be given a 1 month supply of INH and instructed to take one pill each day. Patients in the continuous INH arm will take INH continuously until the end of the study. Depending on when the patient enrolls in the study, the patient could take INH for 1 to 4 years. Each patient will be provided with education on the need to adhere to the protocol and information on potential study drug related toxicity. All patients will be given their first dose of study medication during the enrollment period. Patients in the shorter-course, observed regimens will be given each of their doses in a clinic under the supervision of a study nurse.

At each study encounter, possible toxicity will be assessed via interview. Patients will be followed every 6 months after the completion of preventive therapy until the study closes. Outreach workers will perform home visits to encourage follow-up and determine vital status for any patient who has missed a scheduled follow-up visit. Patients with evidence of active tuberculosis at any follow-up visit will be evaluated and treated appropriately. Patients will be offered a small incentive for fulfilling study requirements. The equivalent of $5 (30 rand) will be paid after successful entry into the trial and at each 6 month visit as compensation for time spent in the study and to cover travel expenses.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Tuberculin test (PPD) positive 5 mm or greater
* Chest x-ray negative for pulmonary tuberculosis

Exclusion Criteria:

* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1148 (Actual)
Dates: Start 2002-09; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Development of confirmed, probable, or possible active pulmonary or extrapulmonary tuberculosis (TB) | 6/2008

SECONDARY OUTCOMES:
Risk of TB and death | 6/2008
rates of adherence, adverse reactions and treatment discontinuation | 6/2008
patterns of antibiotic resistance | 6/2008
clinical and epidemiological factors associated with developing TB | 6/2008

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chaisson, MD, Principal Investigator — Johns Hopkins Medical Institute
Locations (1):
- Chris Hani Baragwanath Hospital, Soweto, South Africa

REFERENCES:
- [Derived] Singh P, Moulton LH, Barnes GL, Gupta A, Msandiwa R, Chaisson RE, Martinson NA. Pregnancy in Women With HIV in a Tuberculosis Preventive Therapy Trial. J Acquir Immune Defic Syndr. 2022 Dec 1;91(4):397-402. doi: 10.1097/QAI.0000000000003078. PMID 36000934
- [Derived] Martinson NA, Barnes GL, Moulton LH, Msandiwa R, Hausler H, Ram M, McIntyre JA, Gray GE, Chaisson RE. New regimens to prevent tuberculosis in adults with HIV infection. N Engl J Med. 2011 Jul 7;365(1):11-20. doi: 10.1056/NEJMoa1005136. PMID 21732833